CLINICAL TRIAL: NCT04166487
Title: Pilot Study of Serial Plasma Genotyping to Guide the Adaptive Treatment of Advanced NSCLC Receiving First-line Pembrolizumab
Brief Title: Plasma-Adapted First-Line Pembro In NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Julia K. Rotow, MD (Other)
Collaborators: Inivata (Industry)
Responsible Party: Sponsor-Investigator, Julia K. Rotow, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-523
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: NSCLC Stage IV; Metastatic Non-Small Cell Lung Cancer
Keywords: NSCLC Stage IV; Metastatic Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Pemetrexed; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Pembrolizumab Cycles 1-2 (Experimental): * For the first two cycles, Pembrolizumab will be administered at a predetermined dose every 3 weeks.
  * InVision plasma draw will take place at Cycle 1 Day 1 and Cycle 2 Day 1, with return of results to the treating oncologist prior to Cycle 3 Day 1.
  * At Cycle 3, patients will be re-registered per the inclusion criteria into 3 arms;
    * PEMBROLIZUMAB Alone
    * PEMBROLIZUMAB + Doublet Chemotherapy
  Interventions: Drug: Pembrolizumab; Diagnostic Test: InVision
- Pembrolizumab Alone, Cycle 3+ (Experimental): - Following imaging assessment at Cycle 3, participants will continue pembrolizumab alone if the following responses are observed:
  * Response of Partial Response/Complete Response
  * Response of Stable Disease with plasma response
  * Response of Progressive Disease without worsening cancer symptoms AND plasma response
  Interventions: Drug: Pembrolizumab
- Pembrolizumab + Doublet Chemotherapy, Cycles 3+ (Experimental): * Following imaging assessment at Cycle 3, participants will receive pembrolizumab in combination with platinum doublet chemotherapy if they have a response of stable disease without plasma response, OR no plasma response and response of progressive disease without worsening cancer systems. Platinum doublet should be histology-appropriate and will be given on-label, per treating oncologist.
  * PEMBROLIZUMAB
  * Chemotherapy multiple agents systemic
    * PEMETREXED
    * CARBOPLATIN
    * PACLITAXEL
  Interventions: Drug: Pembrolizumab; Drug: PEMETREXED; Drug: CARBOPLATIN; Drug: PACLITAXEL

INTERVENTIONS:
Drug: Pembrolizumab — predetermined dose, once per cycle via IV will be administered every 3 weeks, with 21 consecutive days defined as a treatment cycle.
  Other Names: Keytruda®
Drug: PEMETREXED — administered per standard practice, once per cycle via IV will be administered every 3 weeks, with 21 consecutive days defined as a treatment cycle.
  Other Names: Alimta®
  Arms: Pembrolizumab + Doublet Chemotherapy, Cycles 3+
Drug: CARBOPLATIN — administered per standard practice once per cycle via IV will be administered every 3 weeks, with 21 consecutive days defined as a treatment cycle.
  Other Names: Paraplatin ®
  Arms: Pembrolizumab + Doublet Chemotherapy, Cycles 3+
Drug: PACLITAXEL — administered per standard practice once per cycle via IV will be administered every 3 weeks, with 21 consecutive days defined as a treatment cycle.
  Other Names: Taxol®,; Onxal
  Arms: Pembrolizumab + Doublet Chemotherapy, Cycles 3+
Diagnostic Test: InVision — Plasma draw for clinical test performed at C1D1 and C2D1; plasma draw for research testing performed at other timepoints per protocol.
  Arms: Pembrolizumab Cycles 1-2

SUMMARY:
This research study is studying to see if a blood test, collected at different times during the treatment of metastatic non-small lung cancer, can be used to detect early response in patients being treated with pembrolizumab and use that information to determine whether patients should continue treatment with pembrolizumab or switch treatment to pembrolizumab in combination with chemotherapy.

The names of the study drugs involved in this study are:

* Pembrolizumab
* Platinum doublet chemotherapy, which may include the following:

  * Carboplatin and pemetrexed
  * Carboplatin and paclitaxel

The name of the blood test:

- InVision (Inivata, Ltd.)

DETAILED DESCRIPTION:
This is an open label, single institution, prospective pilot study.

The purpose of this research study is to determine if a blood test, collected at different times during treatment, can be used to detect early response in patients being treated with pembrolizumab for lung cancer and use that information to determine whether patients should continue treatment with pembrolizumab or switch treatment to pembrolizumab in combination with chemotherapy.

-The research study procedures include screening for eligibility and study treatment including evaluations approximately every 3 weeks.

The names of the study drugs involved in this study are:

* Pembrolizumab
* Platinum doublet chemotherapy, which may include the following:

  * Carboplatin and pemetrexed
  * Carboplatin and paclitaxel

The name of the blood test:

* InVision- Inivata

  * This blood test that will help study how participants respond to the study treatment. ---
  * Blood will be collected for this test at a few time points, both before and after participants receive treatment on study.
* Participants will be on the research study for up to 12 months.
* It is expected that about 40 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

- Participants must have histologically or cytologically confirmed stage IV NSCLC (AJCC 8th edition).

- Participants must have evaluable disease on imaging per RECIST (measurable disease is not required).

* No prior treatment with a systemic anti-cancer therapy of any kind for the treatment of stage IV NSCLC. Prior definitive chemoradiation for locally advanced disease, or prior adjuvant or neoadjuvant therapy for early stage disease is permitted if completed ≥6 months prior to initiating study treatment.
* Age ≥18 years.
* ECOG performance status 0-2 (see Appendix A)
* Candidate for combination chemoimmunotherapy per physician assessment.
* Participants must have normal organ and marrow function as defined below:

  -- absolute neutrophil count ≥1000/mcL
  * platelets ≥100,000/mcL
  * total bilirubin <1.3 mg/dL
  * creatinine <1.6 mg/dL
* PD-L1 tumor proportion score (TPS) ≥1%, as determined by a CLIA-laboratory.
* The effects of pembrolizumab on the developing human fetus are unknown. For this reason and because immune checkpoint blockade agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of pembrolizumab administration.

  -- NOTE: a pregnancy test will be required at screening for women of childbearing potential.
* Ability to understand and the willingness to sign a written informed consent document.
* Inclusion Criteria for Treatment Continuation at Cycle 3 -- Completion of repeat plasma NGS (InVision) on study, with plasma response defined as ≥50% reduction in plasma ctDNA max AF between C1D1 and C2D1 for patients with high shed [≥0.5% max AF] at C1D1, or continued low shed [<0.5% max AF] for patients with low shed at C1D1.

  * Completion of restaging scans on study, with response determined by central review per RECIST 1.1 criteria
  * For participants continuing pembrolizumab alone:

    * Response of Partial Response or Complete Response at Cycle 3 imaging assessment (as determined by TIMC).

OR --- Response of Stable Disease at Cycle 3 imaging assessment (as determined by TIMC) AND plasma response.

OR

* Response of Progressive Disease at Cycle 3 imaging assessment (as determined by TIMC) without worsening cancer symptoms (as determined by the treating investigator) AND plasma response.

  -- For participants continuing pembrolizumab + doublet chemotherapy:
* Response of Stable Disease at Cycle 3 imaging assessment (as determined by TIMC) AND no plasma response.

OR --- Response of Progressive Disease at Cycle 3 imaging assessment (as determined by TIMC) without worsening cancer symptoms (as determined by the treating investigator) AND no plasma response.

- NOTE: Patients with a response of Progressive Disease at Cycle 3 imaging assessment (as determined by TIMC) with worsening cancer symptoms (as determined by the treating investigator) must come off treatment.

Exclusion Criteria:

* Participants with known sensitizing alterations in EGFR, ALK, ROS1 or BRAF.
* Participants who have had chemotherapy or radiotherapy within 1 week prior to entering the study.
* Participants who are receiving any other investigational agents.
* Participants with uncontrolled brain metastases, leptomeningeal disease, or spinal cord compression. Patients with asymptomatic untreated brain metastases are eligible. Patients with treated CNS disease are eligible if stable disease is clinically confirmed ≥2 weeks after definitive CNS therapy (radiation or surgery), and the patient is not receiving systemic steroids ≥10mg of prednisone equivalent at the time of enrollment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab or other agents used in study.
* Ongoing or active autoimmune disease requiring systemic steroids of ≥10mg of prednisone equivalent or other systemic immunomodulatory agents at the time of enrollment. Type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as psoriasis, vitiligo, and alopecia) not requiring systemic therapy, or conditions not expected to recur in the absence of an external trigger are allowed.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because pembrolizumab is a Pregnancy Category D agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab, breastfeeding should be discontinued if the mother is treated with pembrolizumab. These potential risks may also apply to other agents used in this study.
* Participants with a known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
6-month Progression Free Survival rate | 6 Months
  Kaplan-Meier method

SECONDARY OUTCOMES:
Early Plasma Response | 42 Days (each cycle is 21 days)
  Early plasma response is defined as ≥50% reduction in plasma ctDNA max AF between Cycle 1 Day 1 and Cycle 2 Day 1 for patients with high shed [≥0.5% max AF] at Cycle 1 Day 1, or persistent low shed [<0.5% max AF] for patients with low shed at Cycle 1 Day 1.
Progression Free Survival | he time from registration to the earlier of progression or death due to any cause or 30 Months
  Kaplan-Meier method will be used to estimate event-time distributions and medians for time-to-event data
Overall Survival | time from registration to death from any cause, and patients who are thought to be alive at the time of final analysis will be censored at the last date of contact or 30 months
  Kaplan-Meier method will be used to estimate event-time distributions and medians for time-to-event data
Feasibility-adherence to protocol therapy for 4 cycles | 84 Days (each cycle is 21 days)
  Feasibility is defined as a patient's adherence to protocol therapy for 4 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Julia K Rotow, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber at Steward St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center (DF/BWCC) in clinical affiliation with South Shore Hospital, South Weymouth, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu